CLINICAL TRIAL: NCT03007199
Title: Arrhythmia Genetics in the NEtherlandS
Acronym: AGNES
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Connie Bezzina, Prof. dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: CCMO # 13598
Record Dates: First submitted 2016-12-21; First posted 2017-01-02 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Myocardial Infarction First; Ventricular Fibrillation
MeSH Terms: conditions — Ventricular Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — DNA from blood.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- AGNES Controls: AGNES controls are individuals with a first acute ST-elevation myocardial infarction but without ventricular fibrillation.
- AGNES cases: AGNES cases have ECG- registered ventricular fibrillation occurring before reperfusion therapy for an acute and first ST-elevation myocardial infarction.

SUMMARY:
The AGNES case-control set consists of individuals with a first acute ST-elevation myocardial infarction. AGNES cases have ECG- registered ventricular fibrillation occurring before reperfusion therapy for an acute and first ST-elevation myocardial infarction. AGNES controls are individuals with a first acute ST-elevation myocardial infarction but without ventricular fibrillation. All cases and controls are recruited at seven heart centers in The Netherlands. The investigators' exclude individuals with an actual non-ST-elevation myocardial infarction, prior myocardial infarction, congenital heart defects, known structural heart disease, severe comorbidity, electrolyte disturbances, trauma at presentation, recent surgery, previous coronary artery bypass graft or use of class I and III antiarrhythmic drugs. Individuals who develop ventricular fibrillation during or after percutaneous coronary intervention are not eligible. Furthermore, because early reperfusion limits the opportunity of developing ventricular fibrillation, potential control subjects undergoing percutaneous coronary intervention within 2 h after onset of myocardial ischemia symptoms were not included. This time interval is based on the observation that >90% of cases develop ventricular fibrillation within 2 h after onset of the complaint of symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. First ST elevation myocardial infarction (STEMI)
2. Between 18 and 80 years old

Exclusion Criteria:

1. A grandparent from non-European descent
2. Inborn errors; congenital heart defects.
3. Prior myocardial infarction (either STEMI or non-STEMI)
4. Previous CABG (coronary artery bypass graft)
5. Use of anti-arrhythmic drugs with the exception of beta-blockers, Ca2+-antagonists and lanoxin.
6. Severe current co morbidity (electrolyte disturbances, K+>5.5, K+<3.0 mmol/L, anaemia, trauma, surgery).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases are patients with a first ST-elevation myocardial infarction (STEMI) referred for primary percutaneous intervention (PCI), who develop ventricular fibrillation between the onset of acute myocardial infarction (chest pain, ECG changes) and reperfusion. Reperfusion can either be spontaneous or by PCI.
  Control patients are patients with a first STEMI, referred for PCI who do not develop ventricular fibrillation.
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2010-02; Primary Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Differences in genetic and inflammatory profile between cases and controls. | Immediately upon admission, measures are based on samples taken at admission.
  Differences in genetic profile and inflammatory profile between cases and controls are investigated between the complete cohorts.

SECONDARY OUTCOMES:
Differences in clinical characteristics between cases and controls | Immediately upon admission, measures are based on status at hospital admission.
  Differences in clinical characteristics between cases and controls are investigated between the complete cohorts.

OTHER OUTCOMES:
Previously described risk factors | Immediately upon admission, measures are based on status at hospital admission.
  Clinical characteristics that were previously described as possible risk factors for the development of VF (ventricular Fibrillation) during AMI (acute myocardial infarction): certain ECG characteristics, infarct size, infarct location, extent and localization of coronary disease. Are investigated for differences between cases and controls in the complete cohorts

REFERENCES:
- [Background] Marsman RF, Wilde AA, Bezzina CR. Genetic predisposition for sudden cardiac death in myocardial ischaemia: the Arrhythmia Genetics in the NEtherlandS study. Neth Heart J. 2011 Feb;19(2):96-100. doi: 10.1007/s12471-010-0070-4. Epub 2011 Jan 28. PMID 21461030
- [Result] Bezzina CR, Pazoki R, Bardai A, Marsman RF, de Jong JSSG, Blom MT, Scicluna BP, Jukema JW, Bindraban NR, Lichtner P, Pfeufer A, Bishopric NH, Roden DM, Meitinger T, Chugh SS, Myerburg RJ, Jouven X, Kaab S, Dekker LRC, Tan HL, Tanck MWT, Wilde AAM. Genome-wide association study identifies a susceptibility locus at 21q21 for ventricular fibrillation in acute myocardial infarction. Nat Genet. 2010 Aug;42(8):688-691. doi: 10.1038/ng.623. Epub 2010 Jul 11. PMID 20622880
- [Derived] Gho JMIH, Postema PG, Conijn M, Bruinsma N, de Jong JSSG, Bezzina CR, Wilde AAM, Asselbergs FW. Heart failure following STEMI: a contemporary cohort study of incidence and prognostic factors. Open Heart. 2017 Dec 22;4(2):e000551. doi: 10.1136/openhrt-2016-000551. eCollection 2017. PMID 29296283